CLINICAL TRIAL: NCT05455853
Title: Effect of Bilateral Transcutaneous Tibial Nerve Stimulation on Postpartum Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, walaa salah mohammed ahmed, spechalist of physical therapist at qulin hospital ,kafrelshikh,Egypt ., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.Rec/012/003728
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Exercise; Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral transcutaneous tibial nerve stimulation,exercise and advices (Experimental): •They will receive bilateral transcutaneous tibial nerve stimulation three times per week for 4 weeks, in addition to abdominal muscle training and breathing exercise and bowel care advices.
  Interventions: Other: Experimental: bilateral transcutaneous tibial nerve stimulation,exercise and advices
- Exercises and advices (Experimental): They will perform abdominal muscle training and breathing exercise three times per week, for 4 weeks in addition to bowel care advices.
  Interventions: Other: Experimental: bilateral transcutaneous tibial nerve stimulation,exercise and advices

INTERVENTIONS:
Other: Experimental: bilateral transcutaneous tibial nerve stimulation,exercise and advices — • First group they will receive morning bilateral transcutaneous tibial nerve stimulation, for 30 minutes, three times per week for 4 weeks, in addition to abdominal muscle training and breathing exercise for 15 minutes three times per week, for 4 weeks and bowel care advices.•They will perform abdominal muscle training and breathing exercise, for 15 minutes three times per week, for 4 weeks in addition to bowel care advices.
  Second group•They will perform abdominal muscle training and breathing exercise, for 15 minutes three times per week, for 4 weeks in addition to bowel care advices.
  Other Names: Exercises and advices

SUMMARY:
This study will be conduct to determine the effect of bilateral transcutaneous tibial nerve stimulation on treating postpartum constipation

DETAILED DESCRIPTION:
TTNS was effective in treating constipation .It was believed that re-establishment of normal colonic function may be possible with neuromodulation of sacral nerve stimulation (SNS) that may improve constipation symptoms but it is expensive and invasive . Percutaneous tibial nerve stimulation (PTNS) is an alternative method of neuromodulation that has shown efficacy in constipation and it stimulates L4-S3 nerve roots of sacral plexus that supply the pelvic floor and lower gastrointestinal tract, Transcutaneous tibial nerve stimulation (TTNS) targets the tibial nerve in a similar fashion to PTNS but it is cheaper and does not require needle puncture .There were few studies showed that TTNS has been used and shown to be effective for treating constipation, but till now, there is no previous study illustrating it's effect specifically on postpartum constipation. So, this study will be the first one in this issue.

ELIGIBILITY:
Inclusion Criteria:•Postpartum women, delivered by caesarean section suffering from constipation after delivery.

* Their ages will range from 20 to 35 years old.
* Their body mass index (BMI) will range from 25 to 33 kg/m2.
* All participating women should have at least two criteria of Rome III diagnostic criteria for constipation.

They should stop laxatives intake during treatment program

-

Exclusion Criteria:

Postpartum women will be excluded if they have:

* History of inflammatory bowel disease, and irritable bowel syndrome.
* Endocrine disease or digestive tract disease.
* History of genital prolapse and anal fissure.
* Congental anorectal malformation, stoma in situ.
* Diabtes mellitus and sever distal venous insuffiency.
* Skin eruption at the site of stimulation.
* Implanted pacemaker or defibrillator.
* Metalic implant in lower limb.
* Recent surgery at the lower limb.
* Peripheral neuropathy and neurological disorders. Psychological distress.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The Bristol Stool Form Scale (BSFS) | up to 4 weeks
  It is a formal research tool used to assess stool consistency and intestinal transit rate. It is an ordinal scale used to rate and categorize stool into seven classifications, according to stool consistency It is also useful in evaluating the effectiveness of an intervention for gastrointestinal tract disease and clinical assessment. It helps people to report on stool consistency adequately, thus proving a guide in the diagnosis and treatment of gastrointestinal disorders.It classifies stool into seven categories ranging from hard lumps like nuts stool (type 1) to watery without solid pieces, entirely liquid (type 7). Types 1 and 2 are indicative of constipation, types 3 and 4 are considered normal stool consistency that is easy to defecate, while types 6 and 7 are considered abnormal consistency .
Patient Assessment of Constipation -Symptom Questionnaire (PAC-SYM) | up to 4 weeks
  It is frequently used in clinical trials of constipation, it has emerged as an important tool for assessing the severity of patient-reported symptoms of constipation. It consists of 12-item questionnaire that divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden. Observational data have shown that PAC-SYM questionnaire has internal consistency, test-retest reliability and concurrent validity, and to be responsive to change over time .
Patient Assessment of constipation quality of life questionnaire (PAC-QOL) | up to 4 weeks
  The validated PAC-QOL questionnaire consists of 28 items grouped into 4 subscales ; physical discomfort , psychosocial discomfort, in addition to worries and concerns, and satisfaction, investigating the effects of constipation on the patient's quality of life in the recent 2 weeks. The first three subscale comprise the patient dissatisfaction index (where higher great corresponding to worse quality of life) the satisfaction subscale include 4 items, (where higher great corresponding to improve quality of life .
Rome III criteria: Rome III criteria: Rome III criteria | up to 4 weeks
  It will be used to confirm the diagnosis of constipation for all participating women in both groups A and B to ensure that they will meet the eligibility criteria . All women should have at least two of the following criteria:
  Fewer than three spontaneous bowel movements per week. Straining during at least 25% of defecation attempts. Lumpy or hard stools for at least 25% of defecation attempts. Sensation of anorectal obstruction or blockage for at least 25% of defecation attempts.
  Sensation of incomplete defecation for at least 25% of defecation attempts. Manual maneuvering required to defecate for at least 25% of defecation attempts (e.g., digital evacuation, support of the pelvic floor).
  Loose stools are rarely present without the use of laxatives.

IPD SHARING:
Plan to Share IPD: Yes